CLINICAL TRIAL: NCT04445753
Title: Nurse-Guided Complementary Exercise for Cardiac Function Improvement in Heart Failure: Findings from the Tai-Heart RCT
Brief Title: Tai Chi Exercise in Patients with Heart Failure
Acronym: The Tai-Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Seyma Demir, Research Assist, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AIBU-HSF-SDEMIR-01
Record Dates: First submitted 2020-05-29; First posted 2020-06-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Nursing Caries; Heart Failure; Quality of Life
Keywords: heart failure; quality of life; Tai Chi
MeSH Terms: conditions — Heart Failure | interventions — Aquatic Therapy; Educational Status; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tai Chi program (Experimental): Individuals in the intervention group will perform a 12-week Tai Chi exercise in company with a researcher.Following the warm-up movements (Qi-gong), the training protocol of the Tai Chi movements, which includes the 10-form Yang style, will continue for 12 weeks, with two sessions per week determined by the researchers.The first and second weeks of the exercise protocol will include introducing the Tai Chi philosophy and teaching 10 forms of Yang style to patients. For 12 weeks, individuals will practice 10 forms of Tai Chi exercises with a researcher in each session. Each session will be planned as one hour.
  Interventions: Other: Tai Chi exercise
- Control group (Other): Individuals in the control group will be trained on heart failure. The only attempt to be made to the control group will be education.
  Interventions: Behavioral: Education (control group)

INTERVENTIONS:
Other: Tai Chi exercise — Individuals in the intervention group will perform a 12-week Tai Chi exercise in company with a researcher.Following the warm-up movements (Qi-gong), the training protocol of the Tai Chi movements, which includes the 10-form Yang style, will continue for 12 weeks, with two sessions per week determined by the researchers.The first and second weeks of the exercise protocol will include introducing the Tai Chi philosophy and teaching 10 forms of Yang style to patients. For 12 weeks, individuals will practice 10 forms of Tai Chi exercises with a researcher in each session. Each session will be planned as one hour.
  Arms: Tai Chi program
Behavioral: Education (control group) — Individuals in the control group will also be trained on heart failure, which will be applied to individuals in the intervention group. The only attempt to be made to the control group will be education.
  Arms: Control group

SUMMARY:
Aim: The aim of the present study is to examine with B-type natriuretic peptide (pro-BNP) and echocardiographic parameters and to measure life quality the effects of the 12-week Tai-Chi exercise program on cardiovascular responses in patients with heart failure in Turkey. In addition, four basic research questions have been identified for the purpose of the research:

Methods:Randomized controlled trial will be carried out in the cardiology outpatient clinic in Turkey. The research will include two groups, an intervention (n=23) and a control (n=23). Cardiovascular responses will be measured with Pro-BNP, transthoracic echocardiography and six minutes walking test; Quality of life measurements with Left Ventricular Dysfunction Scale (LVD-36).Tai-Chi exercises will be carried out for a total of 12 weeks, with 2 sessions each week and one hour each session for intervention group. In addition, initially, approximately 45 minutes of heart failure education will be given to both the intervention and control groups.

DETAILED DESCRIPTION:
The aim of the present study is to examine with B-type natriuretic peptide (pro-BNP) and echocardiographic parameters and to measure life quality the effects of the 12-week Tai-Chi exercise program on cardiovascular responses in patients with heart failure in Turkey. In addition, four basic research questions have been identified for the purpose of the research:

1. Methods:

1.1. Design: Randomized controlled trial. 1.2. Setting: The research will be carried out in the cardiology outpatient clinic of Izzet Baysal Training and Research Hospital, Bolu, Turkey.

1.3. Sample: The research will include two groups, an intervention and a control. Power analysis was used to determine the sample size. The sample of 46 (intervention=23, control=23) was sufficient with 0.86 effect size, 95% confidence interval and 80% power. In randomization, closed envelope method will be used.

1.4. Data collecting

1.4.1. Patient Information Form: data regarding demographic and clinical features will be collected.

1.4.2. Cardiovascular responses

1.4.2.1. Pro-BNP Measurements: Pro-BNP levels will be studied from venous blood samples taken for each individual before the study (pre-test) and after 12 weeks (post-test). Blood samples will be taken at least 2 cc into ethylenediamine tetraacetic acid (EDTA) tubes between 8:00 am and 9:00 am after 12 hours of fasting; "Fluorescence immunoassay" method will be used by using "Architect BNP Test" kit.

1.4.2.2. Transthoracic Echocardiography Measurements: In this study, all individuals will receive transthoracic echocardiography twice before the study (pre-test) and after 12 weeks (post-test). Transthoracic echocardiographic examination will be performed with the Philips EPIQ 7 echocardiography device and Philips X5-1 xMatrix 3.5 MHz access probe in the reclining position while resting. Measurements will be made according to the American Echocardiographic Association criteria. In two-dimensional echocardiographic examination, parasternal long / short axis, ventricular wall movements, valve structures and functions will be assessed in apical four chamber views; interventricular septum thickness (IVSd), posterior wall thickness (PWd), left ventricular diastolic and systolic inner diameters (LVIDd / s) will be measured. Left ventricular ejection fraction(LVEF) will be evaluated by M-mod and Simpson methods. Evaluation of diastolic functions will be assessed by transmitral pulse wave and tissue doppler examinations, right ventricular basal and mid diameters will be measured at the end of diastole. Tricuspid annular plane systolic excursion (TAPSE) and S-wave measurements will be performed to evaluate the right ventricular systolic functions. Using the Lacobelli method, epicardial fat thickness measurements will be performed.

1.4.2.3. Six minutes walking test: A starting and ending point (30 meters distance) will be determined and all participants will be asked to walk for 6 minutes between this distance and the total distance they walked will be calculated and recorded. This test will be repeated both at baseline (pretest) and after 12 weeks (posttest).

1.4.2.4. Quality of life measurements: Left Ventricular Dysfunction Scale (LVD-36) is a disease-specific quality of life scale developed by Leary and Jones (2000) to measure the quality of life in patients with heart failure.Scores between 0 and 100 are obtained from the scale and the quality of life decreases as the score obtained increases (Leary and Jones, 2000; Özer & Argon, 2005).In this study, the scale will be administered to individuals at the beginning (pre-test) and 12 weeks later (post-test).

1.4.3. Interventions: Tai-Chi exercises will be carried out for a total of 12 weeks, with 2 sessions each week and one hour each session. In addition, initially, approximately 45 minutes of heart failure education will be given to both the intervention and control groups.

1.4.3.1. Tai-Chi procedure: Tai Chi movements will include the 10-form Yang style following the warm up movements (Qi-gong). The first and second weeks of the exercise protocol will include introducing the Tai Chi philosophy and teaching 10 forms of Yang style to patients. During the 12 weeks, individuals will practice 10 forms of Tai Chi exercises with a researcher in each session.

1.4.3.2.Education protocol on heart failure: The scope of the education will include lifestyle changes, such as nutrition, exercise, weight management, smoking and inappropriate alcohol consumption, which are prepared by the researcher in the light of both literature information and evidence based information in the ESC diagnosis and treatment guide for heart failure. The education method will be reflected on the projection both on verbal expression and computer screen, and will be in the form of visual demonstration with visual materials.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Diagnosed as chronic heart failure by the physician,
* Left ventricular ejection fraction (LVEF) <40%, proven by echocardiography in the past two years,
* New York Heart Association (NYHA) class II and III,
* Sinus rhythm is observed in electrocardiography (ECG),
* Blood pressure values measured before Tai Chi session were 120-160 mmHg for systolic pressure and 80-110 mmHg for diastolic pressure,
* No current anxiolytic or hypnotic treatment,
* Have no psychiatric problems,
* Verbal communication can be established,
* Those who understand and speak Turkish,
* No speech, hearing and vision loss,
* There is no physical limitation that prevents the exercise of standing,
* They have never experienced Tai Chi exercise before,
* Individuals who volunteer to participate in the Tai Chi program during the study

Exclusion Criteria:

* Having unstable angina pectoris, myocardial infarction or major cardiac surgery in the past three months,
* Experiencing dyspnea and exercise tolerance that worsen during rest,
* NYHA class I and IV,
* Type B natriuretic peptide level measured in the last three months is 100 and above,
* Blood pressure values measured before the Tai Chi session are> 120 mmHg or <160 mmHg for systolic pressure and> 80 mmHg or <110 mmHg for diastolic pressure,
* Has hemodynamically significant heart valve disease,
* Having dysrhythmia problems such as ventricular tachyarrhythmia, atrial fibrillation,
* Has a history of cardiac resynchronization therapy in the past 3 months,
* Having chronic diseases such as chronic pulmonary disease and renal failure,
* With uncontrolled diabetes (Hemoglobin A1C ≥ 7 mg / dl),
* Diagnosed with thrombophlebitis,
* Has a history of cardiac transplantation and cardiac device therapy (cardiac pacemaker, implantable cardioverter defibrillator),
* Having physical limitations that prevent standing exercise,
* Do not understand and speak Turkish,
* Speech, hearing and vision loss,
* Individuals who do not volunteer to participate in the Tai Chi program during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-12-21 (Actual)

PRIMARY OUTCOMES:
Pro-BNP levels (pg/ml) | 3-months
  Biomarker to be used to estimate the prognosis of heart failure. The blood taken into 2ml EDTA tubes will be studied.
Transthoracic Echocardiography measurements | 3-months
  Transthoracic echocardiography will be performed to each individual and multiple criteria will be evaluated.In two-dimensional echocardiographic examination, left ventricular ejection fraction will be evaluated by M-mod and Simpson methods.

SECONDARY OUTCOMES:
Six-minute walking test (meter) | 3-months
  It is a widely used test that can be easily applied in evaluating functional capacity and treatment response in individuals with cardiopulmonary disease.During the test, patients are asked to walk as fast as they can without running, and the total distance they walk after 6 minutes is measured.
Quality of life | 3-months
  Left Ventricular Dysfunction Scale is a disease-specific quality of life scale developed by Leary and Jones (2000) to measure the quality of life in patients with heart failure. The questions of the 36-item scale are presented to the patients with two options as true and false. The "true" answers given are added together and the total number of "true" answers found is expressed as a percentage. The minimum and maximum scores that can be obtained from the scale range from 0 to 100, and as the score increases, the quality of life decreases. In this study, a questionnaire will be applied initially and after 12 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma Demir, Res. Assist., Principal Investigator — Bolu Abant Izzet Baysal University, Health Sciences Faculty
Locations (1):
- Bolu Abant Izzet Baysal University Izzet Baysal Training and Research Hospital, Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No